CLINICAL TRIAL: NCT06827314
Title: Pharmacological and Mechanical Support Approaches in the Management of Acute Heart Failure in the Regional Network Model for the Management of Cardiogenic Shock
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: Shock-ER
Record Dates: First submitted 2025-01-09; First posted 2025-02-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2024-12

CONDITIONS: Cardiogenic Shock; Acute Coronary Event
MeSH Terms: conditions — Shock, Cardiogenic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this observational study is to understand and describe the epidemiology of cardiogenic shock in Emilia Romagna with a specific focus on outcome stratified by aetiologies, sex and age. The main outcomes are:

* Incidence of cardiogenic shock (CS) over the total CICU admissions, CS-related in-hospital mortality and length of hospitalization, stratified by aetiologies, sex and age
* Epidemiology of patients admitted with CS, regarding age, gender, etiology and modality of presentation (acute or acute on chronic), echocardiographic and haemodynamic data, treatment strategy with inotropes and/or short-term MCS, cardiac arrest.

This is an observational study without intervention. Patients will be treated according to current clinical practice, according to physician judgment and data sheets of each drug used according to clinical practice.

DETAILED DESCRIPTION:
This is a multicenter observational study with both a retrospective and a prospective cohort.

Study population will include all consecutive patients diagnosed with cardiogenic shock and admitted to the cardiac intensive care unit of the participating centers.

For the patients enrolled at IRCCS Azienda Ospedaliera-Universitaria di Bologna this study will involve a collaboration with UO Cardiologia.

For the retrospective cohort, patients will be selected based on ICD9 discharge codes and included if they fulfill inclusion criteria after review of hospital charts. The retrospective cohort will serve as a historical comparison regarding epidemiology, treatment strategies and survival.

Incidence and workload burden of CICU will be studied comparing the number of CS patients and the total number of admissions in the study period.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years old) admitted to a participating CICU with suspected CS of stage from C to E according to SCAI (Society of cardiovascular intervention)classification of cardiogenic shock.
* Signed informed consent.

Exclusion Criteria:

* CS following cardiac surgery (post-cardiotomy), ● Significant polytrauma or neurological injury.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: For the prospective cohort, study population consists of all consecutive patients diagnosed with CS and admitted to participating CICUs in the Emilia Romagna region. For the prospective cohort patients will be enrolled after study approval and until 31 December 2027.
  Patients will be enrolled upon admission or at the development of CS if already admitted.
  Retrospective data will be collected for five years, starting from January 1st 2018 until the starting date of the study.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-12-06 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Incidence of CS over the total CICU admissions stratified by aetiologies, sex and age. | 5 years
  Incidence
Length of hospitalization, stratified by aetiologies, sex and age. | 5 years
  Days
CS-related in-hospital mortality stratified by aetiologies, sex and age. | 5 years
  Incidence
Epidemiology of patients admitted with CS, regarding age, gender, etiology and modality of presentation (acute or acute on chronic), echocardiographic and haemodynamic data, treatment strategy with inotropes and/or short-term MCS, cardiac arrest. | 5 years
  Demography description
Recovery from cardiogenic shock, defined as improvement to at least SCAI stage B or discharge from CICU to a step-down ward | 5 years
  Recovery from cardiogenic shock
In-hospital survival according to age, etiology, presentation (acute or acute on chronic) and modality of treatment (inotropes or MCS). | 5 years
  In-hospital survival
Rate and reason of unplanned re-hospitalizations within one month after primary discharge | 5 years
  Rate and reason of unplanned re-hospitalizations
Workload burden will be estimated as the percentage of CS admission and the mean duration of CICU stay as compared to other admissions during study period | 5 years
  Workload burden
Rate of adherence to several items and differences between older era (retrospective data) and prospective cohort | 5 years
  Blood counts, ECG, oxygen saturation and respiratory monitoring.

SECONDARY OUTCOMES:
Rate of successful bridge to heart replacement therapy (heart transplant or LVAD implant) in patients potentially eligible (i.e. age < 71 years old) and transferred to IRCCS Policlinico S.Orsola hub center. | 5 years
  Rate of successful bridge to heart replacement therapy
Comparison of survival between patients who underwent HRT as a consequence of CS to elective patients in the study period | 5 years
  Comparison of survival
Description of in-hospital complications such as rate of renal replacement therapy, number of nosocomial infections with therapy and consequent associated mortality. | 5 years
  Description of in-hospital complications
Description of MCS-related complications, including bleeding requiring transfusions, vascular complications including bleeding requiring intervention and limb ischemia. | 5 years
  Description of MCS-related complications

CONTACTS AND LOCATIONS:
Overall Officials: Luciano G Potena, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Bologna, Italy